CLINICAL TRIAL: NCT02446782
Title: A Study to Evaluate the Efficacy and Safety of a Single Dose of an Injectable Antibiotic for the Prophylaxis of Surgical Site and Pleural Space Infection After Medical Thoracoscopy
Brief Title: Efficacy and Safety of Prophylactic Use of an Antibiotic for Medical Thoracoscopy
Acronym: APT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Sahajal Dhooria, Assistant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NK/1816/Res/2440
Record Dates: First submitted 2015-05-09; First posted 2015-05-18 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Pleural Effusion; Pleurisy; Empyema
Keywords: thoracoscopy; pleuroscopy; antibiotic prophylaxis; pleural effusion
MeSH Terms: conditions — Pleural Effusion; Pleurisy; Empyema | interventions — Cefazolin; Clindamycin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cefazolin (Experimental): A single dose of intravenous cefazolin 2 gms will be administered over 10 minutes, dissolved in 100 mL of normal saline between 15 and 30 minutes before the incision. This will be preceded by an intradermal test dose to check for hypersensitivity to the drug. If hypersensitivity is present, the patient will be administered a single dose of intravenous Clindamycin 900 mg.
  Interventions: Drug: Cefazolin
- saline (Placebo Comparator): 100 mL normal saline will be administered intravenously over a period of 10 minutes between 15 and 30 minutes before the incision. An intradermal test dose with normal saline will be administered to this group.
  Interventions: Other: saline

INTERVENTIONS:
Drug: Cefazolin — Cefazolin 2 gm administered in 100 mL normal saline (after skin sensitivity testing) 15-30 minutes before the start of the procedure. Clindamycin 900 mg to be administered if sensitivity detected to cefazolin.
  Other Names: Clindamycin
  Arms: Cefazolin
Other: saline — 100 mL normal saline 15-30 minutes before the start of the procedure
  Arms: saline

SUMMARY:
This is a prospective study to assess the efficacy and safety of a single dose of cefazolin 2g IV for the prophylaxis of surgical site and pleural space infections in patients undergoing medical thoracoscopy.

DETAILED DESCRIPTION:
This is a prospective randomized study to assess the efficacy and safety of a single dose of cefazolin 2g IV for the prophylaxis of surgical site and pleural space infections during medical thoracoscopy.

Consecutive patients who are planned to undergo a medical thoracoscopy (rigid or semirigid) will be enrolled in the study if they satisfy the inclusion and exclusion criteria. One hundred patients will be randomized in 1:1 ratio to receive either of the following: (a) A single dose of intravenous cefazolin 2 gms dissolved in 100 mL of normal saline administered over 10 minutes, between 15 and 30 minutes before the incision, OR (b) 100 mL normal saline administered intravenously over a period of 10 minutes between 15 and 30 minutes before the incision. Thoracoscopy will be performed in the bronchoscopy suite on a spontaneously breathing subject (fasting for 8 h) under conscious sedation (using midazolam, pentazocine, and tramadol) observing complete aseptic precautions.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥12 years
2. Medical thoracoscopy being performed for a pleural effusion for any of the three indications: diagnosis, pleurodesis, or adhesiolysis

Exclusion Criteria:

1. Age ≥80 years
2. Pao2/FIO2< 300;
3. Hemodynamic instability
4. Myocardial infarction or unstable angina in the last 6 wk
5. Lack of pleural space due to adhesions
6. Uncorrected coagulopathy
7. Failure to provide informed consent
8. Patients already taking any antibiotic due to any reason

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Efficacy as assessed by occurrence of wound infection or pleural space infection | 2 months
  (a) Occurrence of wound infection as indicated by development of a purulent discharge from the surgical site or (b) pleural space infection as indicated by development of purulence, fall in sugar levels or gram's stain or culture positivity in the pleural fluid drained by the chest tube on the side of the procedure.

SECONDARY OUTCOMES:
Safety as assessed by adverse effects | 7 days
  Adverse effects arising as a result of the antibiotic administered

CONTACTS AND LOCATIONS:
Locations (1):
- PGIMER, Chandigarh, Chandigarh, India